CLINICAL TRIAL: NCT02468271
Title: Clinimetric Properties of Outcome Measures in Bronchiectasis in the UK
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: Belfast Health and Social Care Trust (Other); South Eastern Health and Social Care Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); NHS Lothian (Other Government); Papworth Hospital NHS Foundation Trust (Other Government); NHS Tayside (Other Government); University Hospital Southampton NHS Foundation Trust (Other); Cardiff and Vale University Health Board (Other Government); Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Stuart Elborn, Professor of Respiratory Medicine/Consultant Physician (Respiratory Medicine), Queen's University, Belfast
Other Study IDs: MR/L011263/1
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Bronchiectasis
Keywords: Clinimetrics; Lung function; Lung clearance index
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma and sputum specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
There is an increasing demand for researchers and regulatory bodies to use robust outcome measures in clinical trials which have evidence of validity, reliability, and responsiveness. There is currently little agreement on the core clinical endpoints that should be used in bronchiectasis. The importance of improving endpoint outcome measurement is well recognised and groups in other conditions have focused on activities to achieve consensus on a core set of outcomes for clinical trials. The Bronch-UK collaboration has explored the current evidence for clinimetric properties of commonly used outcome measures in bronchiectasis (e.g. forced expiratory volume in one second [FEV1], health related quality of life [HRQoL], and pulmonary exacerbations). The results of this extensive rigorous literature review of 68 papers clearly demonstrate that whilst there was good evidence for validity for key outcome measures in bronchiectasis there is little information available on their reliability (during periods of clinical stability) or response to treatment (effect sizes).

The aim of this study is to explore the clinimetric properties of a range of outcome measures, in order to make recommendations for their use in clinical trials in bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is a persistent or progressive condition characterised by dilated thick-walled bronchi. The recent guidelines stipulate that high resolution computerised tomography scan (HRCT) is the radiological investigation of choice to establish the diagnosis of bronchiectasis. The key radiological features of bronchiectasis include bronchial wall dilation (internal lumen diameter greater than accompanying pulmonary artery) which is the characteristic feature of bronchiectasis.

Prevalence of bronchiectasis in most populations is largely inaccurate due to lack of recent studies. United Kingdom (UK) figures indicate prevalence figures of 100/100,000 based on studies undertaken in the 1950's but these did not involve use of high resolution computerised tomography scan for diagnosis. This number is five to ten times higher in people over 55 years of age. The mean age of death is 72 years.

The aetiology for bronchiectasis is variable, however, current data suggests that the most common causes are: post infectious; immunological; congenital; with a proportion also idiopathic.

Bronchiectasis is increasingly being recognised as a major cause of pulmonary morbidity. The signs and symptoms of bronchiectasis include chronic sputum production, shortness of breath and fatigue; all of which contribute to increased morbidity and may progress to respiratory failure and cor pulmonale.

The management of bronchiectasis incorporates an intense regime of prevention and treatment. These often include daily intake of inhaled and nebulised medications, antibiotic therapy, airway clearance, visits to GP and/or respiratory clinics and hospitalisation. The burden of treatment associated with bronchiectasis is therefore significant and is provided at a huge economic cost to the health service. Many of these treatments are provided in the absence of a sound evidence base and so there is a clear need to develop assessment tools for use both in clinical trials and in clinical practice.

There is an increasing demand for researchers and regulatory bodies to use robust outcome measures in clinical trials which have evidence of validity, reliability, and responsiveness. There is currently little agreement on the core clinical endpoints that should be used in bronchiectasis. The importance of improving endpoint outcome measurement is well recognised and groups in other conditions have focused on activities to achieve consensus on a core set of outcomes for clinical trials. The Bronch-UK collaboration has explored the current evidence for clinimetric properties of commonly used outcome measures in bronchiectasis (e.g. forced expiratory volume in one second [FEV1], health related quality of life [HRQoL], and pulmonary exacerbations). The results of this extensive rigorous literature review of 68 papers clearly demonstrate that whilst there was good evidence for validity for key outcome measures in bronchiectasis there is little information available on their reliability (during periods of clinical stability) or response to treatment (effect sizes).

Spirometry is a method of assessing lung function by measuring the volume of air that the patient is able to expel from the lungs after a maximal inspiration. Spirometry is a method for measuring the speed and volume of airflow and is seen as the "gold standard" of testing lung function. Forced expiratory volume in one second (FEV1) in healthy individuals and those with early disease mostly reflects proximal airways, however, the annual rate of change in FEV1 in bronchiectasis is very small and FEV1 is not very responsive to many treatments especially in mild disease. In recent years other measures of lung function are emerging as potential outcome measures in bronchiectasis. The pathological changes in bronchiectasis involve the small airways. Forced expiratory flow between 25 and 75% (FEF25-75) of forced vital capacity (FVC) has been proposed as a sensitive measure of early airways dysfunction. The major barriers to the use of this are that FEF25-75 is very dependent on patient effort, is less reproducible than FEV1 and has poorly defined normal ranges in different age groups. Lung clearance index measured by multiple breath washout (MBW) is a measure of ventilation inhomogeneity and is considered to reflect abnormalities of the smaller airways. Small airway disease caused by inflammation and obstruction leads to ventilation heterogeneity. This will therefore cause an increased number of breaths to remove a tracer gas due to uneven gas mixing and subsequently an increased lung clearance index.

To date, the majority of studies using the lung clearance index have been conducted in cystic fibrosis. These studies have shown that lung clearance index is more sensitive than spirometry at detecting early lung pathology and that it is a sensitive and repeatable clinical endpoint. It has been used as a secondary end-point in the UK cystic fibrosis gene therapy multidose study; Invacaftor study; hypertonic saline study; and, DNase study.

The investigators have conducted some preliminary studies to explore the use of lung clearance index in bronchiectasis and have shown that lung clearance index is repeatable over short periods of time and a more sensitive indicator of computed tomography (CT) scan abnormalities than spirometry in bronchiectasis. Further research is needed to provide data on long term repeatability during periods of stability (noise) and also establish its responsiveness to change (effect size).

Multiple questionnaires including the St Georges Respiratory Questionnaire (SGRQ); Quality of Life - Bronchiectasis (QOL-B) Questionnaire; and, EuroQol 5 Dimension (EQ-5D) have been used to capture the impact of health related quality of life (HRQoL)/patient reported symptoms in bronchiectasis. There is no comparative data to direct choice of the most appropriate questionnaire for use in clinical trials. With respect to individual questionnaires there is also the need to provide data on long term repeatability and reliability.

Aims:

The aim of this study is to explore the clinimetric properties of a range of outcome measures, in order to make recommendations for their use in clinical trials in bronchiectasis. These measures include: lung function (spirometry, lung clearance index); health related quality of life (HRQoL) assessment [St Georges Respiratory Questionnaire (SGRQ); Quality of Life - Bronchiectasis (QOL-B) Questionnaire; EuroQol 5 Dimension (EQ-5D)]; and, blood (white cell count, c-reactive protein) and sputum (microbiology, inflammatory markers) processing.

Specific Objectives:

* To ascertain the relative stability (least noise) of these potential outcome measures in bronchiectasis over a one year timeframe.
* To ascertain the relative effect size of these outcome measures over a pulmonary exacerbation signal interval (greatest signal-to-noise ratio).
* To compare clinimetric properties (reliability, validity and responsiveness to change) of the health related quality of life (HRQoL) questionnaires.

ELIGIBILITY:
Inclusion Criteria

* Proven and documented diagnosis of non-cystic fibrosis idiopathic or post-infectious bronchiectasis by high resolution computerised tomography scan including two or more lobes and dilated airways compatible with bronchiectasis at initial diagnosis.
* Able to perform an acceptable spirometry session - defined as three acceptable or usable efforts per American Thoracic Society/European Respiratory Society criteria.
* Able to perform an acceptable LCI session.
* Participants must be able and willing to read and comprehend written instructions, and comprehend and complete the questionnaires required by the protocol
* After full explanation, participants must have signed an informed consent form indicating that they understand the purpose of and the procedures required for the study and are willing to participate in the study.
* Participant 18 years of age or above.

Exclusion Criteria

* Women who are pregnant, lactating or in whom pregnancy cannot be excluded.
* Anyone who is participating in or has participated in a clinical trial of an investigational medical product (IMP) within four weeks of first visit.
* Any clinical or genetic features of cystic fibrosis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Lung clearance index | 0 months
  Lung clearance index will be measured using the multiple breath inert gas washout (MBW) test. MBW testing measures the functional residual capacity (FRC) and the efficiency with which gas mixes in the lungs. The non-uniformity of ventilation distribution across the lung is often referred to as ventilation inhomogeneity (VI).
  Measurement of lung clearance index in this study will be performed using the Nitrogen Washout, EXHALYZER D, Ecomedics system. Tests will be performed in triplicate and a minimum of 2 tests with coefficient of variation (CV) <5% will be required in order to ensure reliable test.
Spirometry | 0 months
  Spirometry will be performed according to the American Thoracic Society/European Respiratory Society guidelines (Miller et al, 2005). All spirometry manoeuvres will be performed in sitting position whilst wearing nose clips. At least three acceptable manoeuvres will be performed for each time point and the results will meet within-test and between-test criteria for acceptability. A maximum of six manoeuvres will be performed at any time point.
  The following parameters will be recorded as part of the spirometry assessment:
  * FEV1 - Forced expiratory volume in one second (L)
  * FVC - Forced vital capacity (L)
  * FEV1/FVC (ratio)
  * FEF25-75 - Forced expiratory flow between 25 and 75% of forced vital capacity (FVC) (L / sec).
  * Time the participant last administered bronchodilator will be recorded
St Georges Respiratory Questionnaire (SGRQ) | 0 months
  Is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease and has been validated for use in non-cystic fibrosis bronchiectasis (Wilson et al, 1997). It contains 50 items in two parts. Part 1 the symptoms component is concerned with frequency and severity of symptoms (8 items); Part 2 relates to activities that cause or are limited by breathlessness (16 items) and impact components (26 items) (social functioning, psychological disturbances resulting from airways disease). Part 1 contains several scales and Part 2 has dichotomous (true/false) response except the last question which is a 4-point Likert scale. It takes about 10 minutes to complete the questionnaire. The total score ranges from 0-100, with a higher score indicating a poorer health related quality of life. It assesses the impact of symptoms over the preceding four weeks.
Quality of Life-Bronchiectasis (QOL-B) Questionnaire | 0 months
  The Quality of Life-Bronchiectasis (QOL-B) questionnaire is a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for patients with non-cystic fibrosis bronchiectasis. It contains 37 items assessed across eight domains: respiratory symptoms; physical functioning; role; emotional functioning; social functioning; vitality; health perceptions; and, treatment burden. The responses are given in the form of a 4-point Likert scale (except 1 question about sputum colour, which has 6 answer options) with a recall period of 'the last week' (except for the treatment burden and sputum colour questions, which do not specify a recall period). It will take approximately 10-15 minutes to complete this questionnaire. For the outcome, each dimension will be scored separately on a scale of 0 to 100. The questionnaire has demonstrated excellent internal consistency and 2-week test-retest reliability for each scale (Quittner et al, 2014).
EuroQol 5 Dimension (EQ-5D) | 0 months
  EQ-5D is applicable to a wide range of health conditions and treatments. It provides a simple descriptive profile and a single index value for health status. EQ-5D is primarily designed for self-completion by respondents and is ideally suited for use in postal surveys, in clinics and face-to-face interviews. It is cognitively simple, taking only a few minutes to complete.
  The EQ-5D essentially consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Sputum analysis | 0 months
  A spontaneous sputum sample will be collected at each study visit. Where necessary participants will be instructed to perform cycles of two to three forced expiratory techniques (huffs) followed by coughing to enhance expectoration. All sputum expectorated will be collected in a labelled sterile transparent container and immediately frozen at -80°C until shipment to central lab (Queen's University Belfast).
  The first priority for sputum processing will be to conduct molecular analysis for sputum microbiology. In addition, where volume allows, processing for sputum inflammatory markers will also be conducted. Where possible a proportion of the sample will be stored at -80oC for future analysis.
Blood analysis | 0 months
  In total approximately 20mls of blood will be collected from each participant by venepuncture at each visit in accordance with local laboratory procedures in order to analyse white cell count and C-Reactive protein with a 10ml aliquot stored as plasma for inflammatory marker analysis (including but not limited to fibrinogen, TNF alpha, interleukin 6).
Lung clearance index | 4 months
  Lung clearance index will be measured using the multiple breath inert gas washout (MBW) test. MBW testing measures the functional residual capacity (FRC) and the efficiency with which gas mixes in the lungs. The non-uniformity of ventilation distribution across the lung is often referred to as ventilation inhomogeneity (VI).
  Measurement of lung clearance index in this study will be performed using the Nitrogen Washout, EXHALYZER D, Ecomedics system. Tests will be performed in triplicate and a minimum of 2 tests with coefficient of variation (CV) <5% will be required in order to ensure reliable test.
Spirometry | 4 months
  Spirometry will be performed according to the American Thoracic Society/European Respiratory Society guidelines (Miller et al, 2005). All spirometry manoeuvres will be performed in sitting position whilst wearing nose clips. At least three acceptable manoeuvres will be performed for each time point and the results will meet within-test and between-test criteria for acceptability. A maximum of six manoeuvres will be performed at any time point.
  The following parameters will be recorded as part of the spirometry assessment:
  * FEV1 - Forced expiratory volume in one second (L)
  * FVC - Forced vital capacity (L)
  * FEV1/FVC (ratio)
  * FEF25-75 - Forced expiratory flow between 25 and 75% of forced vital capacity (FVC) (L / sec).
  * Time the participant last administered bronchodilator will be recorded
St Georges Respiratory Questionnaire (SGRQ) | 4 months
  Is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease and has been validated for use in non-cystic fibrosis bronchiectasis (Wilson et al, 1997). It contains 50 items in two parts. Part 1 the symptoms component is concerned with frequency and severity of symptoms (8 items); Part 2 relates to activities that cause or are limited by breathlessness (16 items) and impact components (26 items) (social functioning, psychological disturbances resulting from airways disease). Part 1 contains several scales and Part 2 has dichotomous (true/false) response except the last question which is a 4-point Likert scale. It takes about 10 minutes to complete the questionnaire. The total score ranges from 0-100, with a higher score indicating a poorer health related quality of life. It assesses the impact of symptoms over the preceding four weeks.
Quality of Life-Bronchiectasis (QOL-B) Questionnaire | 4 months
  The Quality of Life-Bronchiectasis (QOL-B) questionnaire is a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for patients with non-cystic fibrosis bronchiectasis. It contains 37 items assessed across eight domains: respiratory symptoms; physical functioning; role; emotional functioning; social functioning; vitality; health perceptions; and, treatment burden. The responses are given in the form of a 4-point Likert scale (except 1 question about sputum colour, which has 6 answer options) with a recall period of 'the last week' (except for the treatment burden and sputum colour questions, which do not specify a recall period). It will take approximately 10-15 minutes to complete this questionnaire. For the outcome, each dimension will be scored separately on a scale of 0 to 100. The questionnaire has demonstrated excellent internal consistency and 2-week test-retest reliability for each scale (Quittner et al, 2014).
EuroQol 5 Dimension (EQ-5D) | 4 months
  EQ-5D is applicable to a wide range of health conditions and treatments. It provides a simple descriptive profile and a single index value for health status. EQ-5D is primarily designed for self-completion by respondents and is ideally suited for use in postal surveys, in clinics and face-to-face interviews. It is cognitively simple, taking only a few minutes to complete.
  The EQ-5D essentially consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Sputum analysis | 4 months
  A spontaneous sputum sample will be collected at each study visit. Where necessary participants will be instructed to perform cycles of two to three forced expiratory techniques (huffs) followed by coughing to enhance expectoration. All sputum expectorated will be collected in a labelled sterile transparent container and immediately frozen at -80°C until shipment to central lab (Queen's University Belfast).
  The first priority for sputum processing will be to conduct molecular analysis for sputum microbiology. In addition, where volume allows, processing for sputum inflammatory markers will also be conducted. Where possible a proportion of the sample will be stored at -80oC for future analysis.
Blood analysis | 4 months
  In total approximately 20mls of blood will be collected from each participant by venepuncture at each visit in accordance with local laboratory procedures in order to analyse white cell count and C-Reactive protein with a 10ml aliquot stored as plasma for inflammatory marker analysis (including but not limited to fibrinogen, TNF alpha, interleukin 6).
Lung clearance index | 8 months
  Lung clearance index will be measured using the multiple breath inert gas washout (MBW) test. MBW testing measures the functional residual capacity (FRC) and the efficiency with which gas mixes in the lungs. The non-uniformity of ventilation distribution across the lung is often referred to as ventilation inhomogeneity (VI).
  Measurement of lung clearance index in this study will be performed using the Nitrogen Washout, EXHALYZER D, Ecomedics system. Tests will be performed in triplicate and a minimum of 2 tests with coefficient of variation (CV) <5% will be required in order to ensure reliable test.
Spirometry | 8 months
  Spirometry will be performed according to the American Thoracic Society/European Respiratory Society guidelines (Miller et al, 2005). All spirometry manoeuvres will be performed in sitting position whilst wearing nose clips. At least three acceptable manoeuvres will be performed for each time point and the results will meet within-test and between-test criteria for acceptability. A maximum of six manoeuvres will be performed at any time point.
  The following parameters will be recorded as part of the spirometry assessment:
  * FEV1 - Forced expiratory volume in one second (L)
  * FVC - Forced vital capacity (L)
  * FEV1/FVC (ratio)
  * FEF25-75 - Forced expiratory flow between 25 and 75% of forced vital capacity (FVC) (L / sec).
  * Time the participant last administered bronchodilator will be recorded
St Georges Respiratory Questionnaire (SGRQ) | 8 months
  Is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease and has been validated for use in non-cystic fibrosis bronchiectasis (Wilson et al, 1997). It contains 50 items in two parts. Part 1 the symptoms component is concerned with frequency and severity of symptoms (8 items); Part 2 relates to activities that cause or are limited by breathlessness (16 items) and impact components (26 items) (social functioning, psychological disturbances resulting from airways disease). Part 1 contains several scales and Part 2 has dichotomous (true/false) response except the last question which is a 4-point Likert scale. It takes about 10 minutes to complete the questionnaire. The total score ranges from 0-100, with a higher score indicating a poorer health related quality of life. It assesses the impact of symptoms over the preceding four weeks.
Quality of Life-Bronchiectasis (QOL-B) Questionnaire | 8 months
  The Quality of Life-Bronchiectasis (QOL-B) questionnaire is a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for patients with non-cystic fibrosis bronchiectasis. It contains 37 items assessed across eight domains: respiratory symptoms; physical functioning; role; emotional functioning; social functioning; vitality; health perceptions; and, treatment burden. The responses are given in the form of a 4-point Likert scale (except 1 question about sputum colour, which has 6 answer options) with a recall period of 'the last week' (except for the treatment burden and sputum colour questions, which do not specify a recall period). It will take approximately 10-15 minutes to complete this questionnaire. For the outcome, each dimension will be scored separately on a scale of 0 to 100. The questionnaire has demonstrated excellent internal consistency and 2-week test-retest reliability for each scale (Quittner et al, 2014).
EuroQol 5 Dimension (EQ-5D) | 8 months
  EQ-5D is applicable to a wide range of health conditions and treatments. It provides a simple descriptive profile and a single index value for health status. EQ-5D is primarily designed for self-completion by respondents and is ideally suited for use in postal surveys, in clinics and face-to-face interviews. It is cognitively simple, taking only a few minutes to complete.
  The EQ-5D essentially consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Sputum analysis | 8 months
  A spontaneous sputum sample will be collected at each study visit. Where necessary participants will be instructed to perform cycles of two to three forced expiratory techniques (huffs) followed by coughing to enhance expectoration. All sputum expectorated will be collected in a labelled sterile transparent container and immediately frozen at -80°C until shipment to central lab (Queen's University Belfast).
  The first priority for sputum processing will be to conduct molecular analysis for sputum microbiology. In addition, where volume allows, processing for sputum inflammatory markers will also be conducted. Where possible a proportion of the sample will be stored at -80oC for future analysis.
Blood analysis | 8 months
  In total approximately 20mls of blood will be collected from each participant by venepuncture at each visit in accordance with local laboratory procedures in order to analyse white cell count and C-Reactive protein with a 10ml aliquot stored as plasma for inflammatory marker analysis (including but not limited to fibrinogen, TNF alpha, interleukin 6).
Lung clearance index | 12 months
  Lung clearance index will be measured using the multiple breath inert gas washout (MBW) test. MBW testing measures the functional residual capacity (FRC) and the efficiency with which gas mixes in the lungs. The non-uniformity of ventilation distribution across the lung is often referred to as ventilation inhomogeneity (VI).
  Measurement of lung clearance index in this study will be performed using the Nitrogen Washout, EXHALYZER D, Ecomedics system. Tests will be performed in triplicate and a minimum of 2 tests with coefficient of variation (CV) <5% will be required in order to ensure reliable test.
Spirometry | 12 months
  Spirometry will be performed according to the American Thoracic Society/European Respiratory Society guidelines (Miller et al, 2005). All spirometry manoeuvres will be performed in sitting position whilst wearing nose clips. At least three acceptable manoeuvres will be performed for each time point and the results will meet within-test and between-test criteria for acceptability. A maximum of six manoeuvres will be performed at any time point.
  The following parameters will be recorded as part of the spirometry assessment:
  * FEV1 - Forced expiratory volume in one second (L)
  * FVC - Forced vital capacity (L)
  * FEV1/FVC (ratio)
  * FEF25-75 - Forced expiratory flow between 25 and 75% of forced vital capacity (FVC) (L / sec).
  * Time the participant last administered bronchodilator will be recorded
St Georges Respiratory Questionnaire (SGRQ) | 12 months
  Is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease and has been validated for use in non-cystic fibrosis bronchiectasis (Wilson et al, 1997). It contains 50 items in two parts. Part 1 the symptoms component is concerned with frequency and severity of symptoms (8 items); Part 2 relates to activities that cause or are limited by breathlessness (16 items) and impact components (26 items) (social functioning, psychological disturbances resulting from airways disease). Part 1 contains several scales and Part 2 has dichotomous (true/false) response except the last question which is a 4-point Likert scale. It takes about 10 minutes to complete the questionnaire. The total score ranges from 0-100, with a higher score indicating a poorer health related quality of life. It assesses the impact of symptoms over the preceding four weeks.
Quality of Life-Bronchiectasis (QOL-B) Questionnaire | 12 months
  The Quality of Life-Bronchiectasis (QOL-B) questionnaire is a self-administered, patient-reported outcome measure assessing symptoms, functioning and health-related quality of life for patients with non-cystic fibrosis bronchiectasis. It contains 37 items assessed across eight domains: respiratory symptoms; physical functioning; role; emotional functioning; social functioning; vitality; health perceptions; and, treatment burden. The responses are given in the form of a 4-point Likert scale (except 1 question about sputum colour, which has 6 answer options) with a recall period of 'the last week' (except for the treatment burden and sputum colour questions, which do not specify a recall period). It will take approximately 10-15 minutes to complete this questionnaire. For the outcome, each dimension will be scored separately on a scale of 0 to 100. The questionnaire has demonstrated excellent internal consistency and 2-week test-retest reliability for each scale (Quittner et al, 2014).
EuroQol 5 Dimension (EQ-5D) | 12 months
  EQ-5D is applicable to a wide range of health conditions and treatments. It provides a simple descriptive profile and a single index value for health status. EQ-5D is primarily designed for self-completion by respondents and is ideally suited for use in postal surveys, in clinics and face-to-face interviews. It is cognitively simple, taking only a few minutes to complete.
  The EQ-5D essentially consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Sputum analysis | 12 months
  A spontaneous sputum sample will be collected at each study visit. Where necessary participants will be instructed to perform cycles of two to three forced expiratory techniques (huffs) followed by coughing to enhance expectoration. All sputum expectorated will be collected in a labelled sterile transparent container and immediately frozen at -80°C until shipment to central lab (Queen's University Belfast).
  The first priority for sputum processing will be to conduct molecular analysis for sputum microbiology. In addition, where volume allows, processing for sputum inflammatory markers will also be conducted. Where possible a proportion of the sample will be stored at -80oC for future analysis.
Blood analysis | 12 months
  In total approximately 20mls of blood will be collected from each participant by venepuncture at each visit in accordance with local laboratory procedures in order to analyse white cell count and C-Reactive protein with a 10ml aliquot stored as plasma for inflammatory marker analysis (including but not limited to fibrinogen, TNF alpha, interleukin 6).

CONTACTS AND LOCATIONS:
Overall Officials: Judy M Bradley, PhD, Principal Investigator — Belfast Health and Social Care Trust; Michael Loebinger, MD, Principal Investigator — Royal Brompton and Harefield Trust; Stephen Rowan, MD, Principal Investigator — South Eastern Health and Social Care Trust; Adam Hill, MD, Principal Investigator — NHS Lothian; Charles Haworth, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust; James Chalmers, MD, Principal Investigator — NHS Tayside; Mary Carroll, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust; James Duckers, MD, Principal Investigator — Cardiff and Vale University Health Board
Locations (7):
- United Kingdom (7):
  - Papworth Hospital, NHS Foundation Trust, Cambridge, England
  - Royal Brompton and Harefield Trust, London, England
  - University Hospital Southampton, NHS Foundation Trust, Southampton, England
  - Belfast Health and Social Care Trust, Belfast, Northern Ireland
  - NHS Tayside, Dundee, Scotland
  - NHS Lothian, Edinburgh, Scotland
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster

REFERENCES:
- [Derived] O'Neill K, Lakshmipathy GR, Neely C, Cosgrove D, Ferguson K, McLeese R, Hill AT, Loebinger MR, Carroll M, Chalmers JD, Gatheral T, Johnson C, De Soyza A, Hurst JR, Bradbury I, Elborn JS, Bradley JM. Multiple-Breath Washout Outcome Measures in Adults with Bronchiectasis. Ann Am Thorac Soc. 2022 Sep;19(9):1489-1497. doi: 10.1513/AnnalsATS.202006-584OC. PMID 35451922